CLINICAL TRIAL: NCT05980442
Title: Randomized, Controlled, Single Center Observational Study to Compare the Safety and Performance of Navigation-assisted OrthoPilot® Elite and Robotic-assisted MAKO® Total Knee Arthroplasty
Brief Title: Comparative Study of Navigation-assisted OrthoPilot® Elite and Robotic-assisted MAKO® Total Knee Arthroplasty
Acronym: ORMAK
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-23032
Record Dates: First submitted 2023-07-19; First posted 2023-08-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis, Knee; Joint Diseases; Rheumatoid Arthritis of Knee; Posttraumatic Arthropathy
Keywords: computer assisted orthopedic surgery; robotic assisted orthopedic surgery; orthopedic navigation; total knee arthroplasty; total knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OrthoPilot® Elite: navigated / computer assisted total knee replacement surgery
  Interventions: Device: Navigated total knee arthroplasty
- MAKO: robot assisted total knee replacement surgery
  Interventions: Device: Robot assisted total knee arthroplasty

INTERVENTIONS:
Device: Navigated total knee arthroplasty — Total knee arthroplasty with Columbus® total knee endoprosthesis using the OrthoPilot® Elite navigation system
  Other Names: Columbus® total knee endoprosthesis
  Groups: OrthoPilot® Elite
Device: Robot assisted total knee arthroplasty — Total knee arthroplasty with Triathlon® total knee endoprosthesis using the MAKO® robot system
  Other Names: Triathlon® total knee endoprosthesis
  Groups: MAKO

SUMMARY:
Randomized, controlled, single center observational study to compare the safety and performance of navigation-assisted OrthoPilot Elite and robotic-assisted MAKO total knee arthroplasty (TKA). The aim of the study is the comparison of the clinical outcome between navigated and robotic-assisted TKA. The hypothesis of the study is that both treatments achieve similar results regarding functional and clinical aspects.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a TKA with a fixed-bearing total knee endoprosthesis
* Written informed consent for participating in the clinical study

Exclusion Criteria:

* Patient age <18 years and >90 years
* Patient not willing to participate at the follow-up
* Pregnancy
* retropatellar arthrosis requiring patella resurfacing
* American Society of Anaesthesiologists (ASA) Classification >3

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 90 years of age having indication for a fixed-bearing total knee endoprosthesis, without retropatellar arthrosis requiring patella resurfacing
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome of the Knee Surgery measured by the Knee Society Score (KSS) (functional component) | one year postoperatively
  Functional result one year postoperatively measured with the functional component of the Knee Society Score (KSS). The KSS is an examiner-administrated standard clinical evaluation tool reporting results for patients undergoing TKA.
  It separates findings in the operated knee (kKSS) score from findings related to the patient's function (fKSS), which might be affected by co-morbidities. The two sub-scores are reported separately ranging from 0 points (worst result) to 100 points (best results), as well as summarized score, total KSS. Final grading of total KSS results Scores of 160 to 200 will be rated as excellent, 140 to 159 as good, 120 to 139 as fair, and less than 120 as poor.

SECONDARY OUTCOMES:
Survival of the implant components | one year postoperatively
  Kaplan-Meier Analysis is a standard statistical method to describe the survival of human subjects or medical products over a defined time period. The revision-free survival rate is the performance indicator of the product under investigation and confirms the clinical outcome of the knee prosthesis. Information on survival of the implant will be collected.
Clinical outcome of the Knee Surgery measured by the Knee Society Score (KSS) (clinical component) | one year postoperatively
  Functional result one year postoperatively measured with the functional component of the Knee Society Score (KSS). The KSS is an examiner-administrated standard clinical evaluation tool reporting results for patients undergoing TKA.
  It separates findings in the operated knee (kKSS) score from findings related to the patient's function (fKSS), which might be affected by co-morbidities. The two sub-scores are reported separately ranging from 0 points (worst result) to 100 points (best results), as well as summarized score, total KSS. Final grading of total KSS results Scores of 160 to 200 will be rated as excellent, 140 to 159 as good, 120 to 139 as fair, and less than 120 as poor.
Quality of Life [EQ-5D-5L] | one year postoperatively
  EQ-5D is a standardized 5-dimension (5D) 5-level (5L) measure of the health status and is developed by the EuroQol Group in order to have a simple and generic measure for clinical and economic assessment. Instructions for the user are directly included into the questionnaire and it consists of two pages. One cover five different dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and the other one the EQ visual Analogue Scale (EQ-VAS). The VAS scale records the self rated health status of the patient from the level "the worst health you can imagine" to "the best health you can imagine".
Anterior knee pain | one year postoperatively
  Anterior knee pain is used to evaluate the performance of the implantation and the implant itself. Rating is classified according to the description of Waters and Bentley in four dimensions: 0 (no pain), I (Mild pain that does not intrude on daily activities), II (Moderate pain that is a nuisance; patient not considering further surgery), III (Severe pain; Patient considering further surgery). The scoring is according to Feller et al. 0, 5, 10 and 15 points, respectively.
Comparison of Radiographic alignment | one year postoperatively
  Alignment (femoral-knee baseline angle, tibial-knee baseline angle, femoral-tibial angle (mechanical))
Comparison of Radiographic status | one year postoperatively
  potential presence of radiolucency at the interface between implant and bone on femoral and tibial components will be analyzed
(Serious) Adverse Events | During the course of the study up to one year postoperatively
  During the course of the study, any upcoming intra- or postoperative (serious) adverse device events or effects ((S)AE) related or not related to the product under investigation, will be documented. The total number of (S)AEs will be summarized and further evaluated by the sponsor and reported according to local legislation and necessity. Recorded complications will be categorized and analyzed in order to assess the safety of the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joachim Riesner, PD Dr. med., Principal Investigator — Bundeswehr Krankenhaus Ulm
Locations (1):
- Bundeswehr Krankenhaus Ulm, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No